CLINICAL TRIAL: NCT02382679
Title: Vitamin Therapy in Concussion Management: A Randomized Control Trial
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was halted prematurely due to enrollment issues
Sponsor: Thomas Jefferson University (Other)
Collaborators: Rothman Institute Orthopaedics (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14D.529
Record Dates: First submitted 2015-03-03; First posted 2015-03-09 (Estimated); Last update posted 2022-04-13 (Actual); Status verified 2022-04

CONDITIONS: Concussion
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Placebo (Placebo Comparator): Non-nutritional non-immunogenic non-allergic oil-based capsule with same appearance, weight and density of active experimental vitamin.
  Interventions: Dietary Supplement: Placebo
- Experimental: Vitamin Mixture (Experimental): Vitamin coenzyme Q10, magnesium, riboflavin and omega-3-fatty acid combination.
  Interventions: Dietary Supplement: Experimental: Vitamin Mixture

INTERVENTIONS:
Dietary Supplement: Experimental: Vitamin Mixture — Vitamins: B2 (riboflavin), magnesium, co-enzyme Q10, Omega 3 fatty acids
  Arms: Experimental: Vitamin Mixture
Dietary Supplement: Placebo — Non-nutritional non-immunogenic non-allergic oil-based capsule with same appearance, weight and density of active experimental vitamin.
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the efficacy of vitamin therapy in concussion when compared to placebo with respect to multiple endpoints including symptom severity, cognitive performance on computer based neuropsychological testing, post-concussion balance assessment, and post-concussion vestibular-oculomotor function.

DETAILED DESCRIPTION:
To date, very little data exists on the use of vitamin supplementation to aid in the recovery of concussion. Data previously published shows potential benefit of certain vitamins in the management of migraine headache. These vitamins, Vitamin B2 (Riboflavin), Magnesium, Co-Enzyme Q-10, and Omega-3 fatty acids, at dosages described in the literature, are being used based on the migraine literature findings and anecdotal evidence to help treat complaints of headache in concussion management.

ELIGIBILITY:
Inclusion Criteria:

* Subjects ages 11-22
* Concussion within 7 days of enrollment
* Presenting for treatment at Rothman Institute or Jefferson Concussion Center

Exclusion Criteria:

* Subjects with recent prior concussion within the past 30 days
* Subjects with a history of moderate to severe TBI requiring hospitalization or resulting in prolonged symptoms (>3weeks).
* Subjects with known neurologic diagnosis associated with impaired cognitive function other that Attention Deficit Hyperactive Disorder or Attention Deficit Disorder.
* Subjects with know allergy to algae, omega-3 fatty acid, or any component of the formulation.
* Subjects currently requiring anticoagulants (ie- Warfarin), anti-platelets (ie- Aspirin, Plavix), or any non-steroidal anti-inflammatory drugs (ie- Ibuprofen, Naprosyn).
* Subjects with known liver pathology or significantly elevated liver function tests (greater than 3 X normal).
* Subjects with a current lower extremity injury that will affect postural stability testing.
* Subjects who are pregnant and/or breast feeding.

Ages: 11 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
PCSI: Post-Concussion Symptom Inventory | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Steve Stache, MD, Principal Investigator — Rothman Institute; Mijail Serruya, MD, PhD, Principal Investigator — Thomas Jefferson University; Robert Franks, DO, Principal Investigator — Rothman Institute; Jeremy Close, MD, Principal Investigator — Thomas Jefferson University

REFERENCES:
- [Background] Sandor PS, Di Clemente L, Coppola G, Saenger U, Fumal A, Magis D, Seidel L, Agosti RM, Schoenen J. Efficacy of coenzyme Q10 in migraine prophylaxis: a randomized controlled trial. Neurology. 2005 Feb 22;64(4):713-5. doi: 10.1212/01.WNL.0000151975.03598.ED. PMID 15728298
- [Background] Schiapparelli P, Allais G, Castagnoli Gabellari I, Rolando S, Terzi MG, Benedetto C. Non-pharmacological approach to migraine prophylaxis: part II. Neurol Sci. 2010 Jun;31 Suppl 1:S137-9. doi: 10.1007/s10072-010-0307-4. PMID 20464605
- [Background] Esposito M, Carotenuto M. Ginkgolide B complex efficacy for brief prophylaxis of migraine in school-aged children: an open-label study. Neurol Sci. 2011 Feb;32(1):79-81. doi: 10.1007/s10072-010-0411-5. Epub 2010 Sep 25. PMID 20872034
- [Background] Bianchi A, Salomone S, Caraci F, Pizza V, Bernardini R, D'Amato CC. Role of magnesium, coenzyme Q10, riboflavin, and vitamin B12 in migraine prophylaxis. Vitam Horm. 2004;69:297-312. doi: 10.1016/S0083-6729(04)69011-X. PMID 15196887
- [Background] Lewis D, Ashwal S, Hershey A, Hirtz D, Yonker M, Silberstein S; American Academy of Neurology Quality Standards Subcommittee; Practice Committee of the Child Neurology Society. Practice parameter: pharmacological treatment of migraine headache in children and adolescents [RETIRED]: report of the American Academy of Neurology Quality Standards Subcommittee and the Practice Committee of the Child Neurology Society. Neurology. 2004 Dec 28;63(12):2215-24. doi: 10.1212/01.wnl.0000147332.41993.90. PMID 15623677